CLINICAL TRIAL: NCT02558231
Title: The Efficacy and Safety of Initial Triple Versus Initial Dual Oral Combination Therapy in Patients With Newly Diagnosed Pulmonary Arterial Hypertension: A Multi-center, Double-blind, Placebo-controlled, Phase 3b Study
Brief Title: The Efficacy and Safety of Initial Triple Versus Initial Dual Oral Combination Therapy in Patients With Newly Diagnosed Pulmonary Arterial Hypertension
Acronym: TRITON
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-065A308
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Results first posted 2020-09-11 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan; Tadalafil; selexipag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triple oral combination treatment (Experimental): Macitentan, tadalafil, and selexipag
  Interventions: Drug: Macitentan; Drug: Tadalafil; Drug: Selexipag
- Dual oral combination treatment (Placebo Comparator): Macitentan, tadalafil, and placebo
  Interventions: Drug: Macitentan; Drug: Tadalafil

INTERVENTIONS:
Drug: Macitentan — Used open-label in both arms, 10 mg tablet, 1 tablet u.i.d.
Drug: Tadalafil — Used open-label in both arms, 20 mg tablet, 1-2 tablets u.i.d.
Drug: Selexipag — Used double-blind in the triple oral treatment arm, 200 microgram tablet, 1-8 tablets b.i.d.
  Arms: Triple oral combination treatment

SUMMARY:
The objective of this clinical trial is to compare the efficacy and safety of an initial triple oral treatment regimen (macitentan, tadalafil, selexipag) versus an initial dual oral treatment regimen (macitentan, tadalafil, placebo) in newly diagnosed, treatment-naïve patients with pulmonary arterial hypertension.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to any study-mandated procedure.
2. Male or female ≥ 18 and ≤ 75 years of age at screening.
3. Initial PAH diagnosis < 6 months prior to enrollment.
4. RHC performed between Day -28 and Day 1, meeting all the following criteria:

   * Mean pulmonary artery pressure (mPAP) ≥ 25 mmHg.
   * Pulmonary artery wedge pressure or left ventricular end-diastolic pressure ≤ 15 mmHg.
   * PVR ≥ 480 dyn•sec/cm5 (≥ 6 Wood Units).
   * Negative vasoreactivity test mandatory in idiopathic, heritable, and drug/toxin induced PAH (at this or a previous RHC).
5. Symptomatic PAH belonging to one of the following subgroups:

   * Idiopathic.
   * Heritable.
   * Drug or toxin induced.
   * Associated with one of the following: connective tissue disease; HIV infection; congenital heart disease.
6. 6-minute walk distance (6MWD) ≥ 50 m at screening.
7. Women of childbearing potential must not be pregnant, must perform regular pregnancy tests, and use reliable contraception.

Exclusion Criteria:

1. Any PAH-specific drug therapy at any time.
2. Cardio pulmonary rehabilitation program based on exercise (planned, or started ≤ 12 weeks prior to Day 1).
3. Body mass index (BMI) > 40 kg/m2 at screening.
4. Presence of three or more of the following risk factors for heart failure with preserved ejection fraction at screening:

   * BMI > 30 kg/m2.
   * Diabetes mellitus of any type.
   * Essential hypertension.
   * Coronary artery disease, i.e., any of the following:

     * History of stable angina or
     * More than 50% stenosis in a coronary artery (by coronary angiography) or
     * History of myocardial infarction or
     * History of or planned coronary artery bypass grafting and/or coronary artery stenting.
5. Acute myocardial infarction ≤ 12 weeks prior to screening.
6. Stroke ≤ 12 weeks prior to screening.
7. Known permanent atrial fibrillation.
8. SBP < 90 mmHg at screening or Day 1.
9. Ongoing or planned treatment with organic nitrates and/or doxazosin.
10. Presence of one or more of the following signs of relevant lung disease at any time up to screening:

    * Diffusing capacity of the lung for carbon monoxide (DLCO) < 40% of predicted (eligible only if no or mild interstitial lung disease on computed tomography).
    * Forced vital capacity (FVC) < 60% of predicted.
    * Forced expiratory volume in one second (FEV1) < 60% of predicted.
11. Known or suspected pulmonary veno-occlusive disease (PVOD).
12. Documented severe hepatic impairment (with or without cirrhosis) according to National Cancer Institute organ dysfunction working group criteria, defined as total bilirubin > 3 × upper limit of the normal range (ULN) accompanied by aspartate aminotransferase (AST) > ULN (assessed by central laboratory at screening); and/or Child-Pugh Class C.
13. Serum AST and/or alanine aminotransferase (ALT) > 3 × ULN (assessed by central laboratory at screening).
14. Severe renal impairment (estimated creatinine clearance ≤ 30 mL/min/1.73 m2) assessed by central laboratory at screening.
15. Ongoing or planned dialysis.
16. Hemoglobin < 100 g/L assessed by central laboratory at screening.
17. Known or suspected uncontrolled thyroid disease (hypo- or hyperthyroidism).
18. Loss of vision in one or both eyes because of non-arteritic ischemic optic neuropathy (NAION).
19. Treatment with strong inducers of cytochrome P450 3A4 (CYP3A4; e.g., carbamazepine, rifampin, rifampicin, rifabutin, rifapentin, phenobarbital, phenytoin, and St. John's wort) ≤ 28 days prior to Day 1.
20. Treatment with strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, nefazodone, ritonavir, and saquinavir) and/or strong inhibitors of CYP2C8 (e.g., gemfibrozil) ≤ 28 days prior to Day 1.
21. Treatment with another investigational drug (planned, or taken ≤ 12 weeks prior to Day 1).
22. Hypersensitivity to any of the 3 study treatments or any excipient of their formulations.
23. Pregnancy, breastfeeding, or intention to become pregnant during the study.
24. Concomitant life-threatening disease with a life expectancy < 12 months.
25. Alcohol abuse.
26. Any factor or condition likely to affect protocol compliance of the subject, as judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (58):
- United States (20):
  - Arizona Pulmonary Specialists, LTD, Phoenix, Arizona
  - UCSD Health Sciences, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Piedmont Pulmonary and Critical Care Research, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - LSU Health Sciences Center, New Orleans, Louisiana
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, Saint Louis, Michigan
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - The Christ Hospital, Cincinnati, Ohio
  - Allegheny General Hospital of Research, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
- Australia (2):
  - Royal Prince Albert Hospital, Camperdown, New South Wales
  - St. Vincents Hospital Sydney, Darlinghurst, New South Wales
- Austria (3):
  - LKH -Universität Klinkum Graz, Graz
  - Krankenhaus der Elisabethinen Linz, Linz
  - AKH Wien, Vienna
- Belgium (2):
  - Hôpital Erasme, Brussels
  - UZ Leuven - Campus Gasthuisberg, Leuven
- Canada (7):
  - Vancouver General Hospital, Vancouver, British Columbia
  - London Health Sciences Centre - Victoria Hospital, London, Ontario
  - University of Toronto, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec
  - University of Calgary, Calgary
  - University of Ottawa Heart Institute, Ottawa
- Denmark (2):
  - Aarhus University Hospital Skejby, Aarhus
  - Rigshospitalet Copenhagen, Copenhagen
- CHU de Bicêtre, Le Kremlin-Bicêtre, France
- Germany (7):
  - Universitätsklinikum Köln, Cologne
  - Unversitätsklinikum Carl Gustav Carus, Dresden
  - Universitätsklinikum Giessen, Giessen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Regensburg, Regensburg
- Mater Misericordiae University Hospital, Dublin, Ireland
- Ospedale Sant'Orsola, Bologna, Italy
- Netherlands (2):
  - VUmc Amsterdam, Amsterdam
  - Maastricht University Medical Center, Maastricht
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital 12 de Octubre, Madrid
- Sweden (3):
  - Skånes universitetssjukhus Lund, Lund
  - Norrlands universitetssjukhus, Umeå
  - Kardiologkliniken, Uppsala
- Universiätsspital Zürich, Zurich, Switzerland
- United Kingdom (4):
  - Golden Jubilee National Hospital, Clydebank
  - The Royal Free Hospital, London
  - Royal Brompton Hospital, London
  - Hammersmith Hospital, London

REFERENCES:
- [Derived] Chin KM, Sitbon O, Doelberg M, Feldman J, Gibbs JSR, Grunig E, Hoeper MM, Martin N, Mathai SC, McLaughlin VV, Perchenet L, Poch D, Saggar R, Simonneau G, Galie N. Three- Versus Two-Drug Therapy for Patients With Newly Diagnosed Pulmonary Arterial Hypertension. J Am Coll Cardiol. 2021 Oct 5;78(14):1393-1403. doi: 10.1016/j.jacc.2021.07.057. PMID 34593120

RESULTS

PARTICIPANT FLOW:
Groups:
- Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag): Participants received macitentan oral tablet, 10 milligrams (mg) once daily and tadalafil oral tablet, 20 mg, once daily from Day 1 up to End of treatment (10 months after last participant was enrolled). Tadalafil was up-titrated from 20 mg to 40 mg on Day 8. In addition, participants received selexipag oral tablet at a starting dose of 200 micrograms (mcg), twice daily from Day 15 up-titrated to a maximum of 1600 mcg, up to End of treatment (10 months after last participant was enrolled).
- Double Oral Therapy (Macitentan, Tadalafil, and Placebo): Participants received macitentan oral tablet, 10 mg once daily and tadalafil oral tablet, 20 once daily from Day 1 up to End of treatment (10 months after last participant was enrolled). Tadalafil was up-titrated from 20 mg to 40 mg on Day 8. In addition, participants received placebo matching to selexipag oral tablet, at a starting dose of 200 micrograms (mcg), twice daily from Day 15 and dose up-titrated to a maximum of 1600 mcg, up to End of treatment (10 months after last participant was enrolled).
Period: Overall Study
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo)
Started | 123 | 124
Treated | 123 | 123
Completed | 98 | 98
Not Completed | 25 | 26
Not completed — Death | 4 | 12
Not completed — Lost to Follow-up | 7 | 4
Not completed — Withdrawal by Subject | 7 | 4
Not completed — Physician Decision | 7 | 5
Not completed — Sponsor Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) includes all randomized participants.
Units Other Than Participants: Number
Groups:
- Total: Total of all reporting groups
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo) | Total
Number analyzed (Participants) | 123 | 124 | 247
Number analyzed (Number) | 123 | 124 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (13.48) | 51.6 (13.92) | 51.9 (13.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 94 | 187
  Male | 30 | 30 | 60
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 20
  Not Hispanic or Latino | 106 | 108 | 214
  Unknown or Not Reported | 7 | 6 | 13
Race/Ethnicity, Customized [Number; unit: participants]
  Black or African American | 5 | 5 | 10
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Asian | 7 | 3 | 10
  White | 102 | 108 | 210
  Other | 3 | 3 | 6
  Unknown or Not Reported | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  AUSTRALIA | 2 | 2 | 4
  AUSTRIA | 9 | 5 | 14
  BELGIUM | 2 | 5 | 7
  CANADA | 11 | 14 | 25
  DENMARK | 3 | 2 | 5
  FRANCE | 4 | 5 | 9
  GERMANY | 13 | 23 | 36
  IRELAND | 1 | 0 | 1
  ITALY | 5 | 6 | 11
  NETHERLANDS | 2 | 2 | 4
  SPAIN | 2 | 1 | 3
  SWEDEN | 7 | 0 | 7
  SWITZERLAND | 1 | 1 | 2
  UNITED KINGDOM | 3 | 2 | 5
  UNITED STATES | 58 | 56 | 114

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in Pulmonary Vascular Resistance (PVR)
Description: Change from baseline to Week 26 in PVR was expressed as the ratio of Week 26 to baseline PVR value (Week 26 divided by baseline) using re-calculated PVR. PVR was determined by right heart catheterization (RHC). A geometric least square mean ratio of Week 26 to baseline PVR less than (<) 1 corresponds to a reduction in PVR from baseline. Missing values were imputed using a last observation carried forward (LOCF) approach.
Time Frame: Baseline, Week 26
Population: Full analysis set (FAS) included all randomized participants.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo)
Number analyzed (Participants) | 123 | 124
ratio | 0.46 [0.422 to 0.503] | 0.48 [0.441 to 0.526]
Statistical Analysis 1: Comparison: Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) vs Double Oral Therapy (Macitentan, Tadalafil, and Placebo); Test type: Superiority; p = 0.4239, ANCOVA; Ratio of geometric Least Square mean = 0.96, 95% CI 2-sided [0.86 to 1.07]

2. Secondary Outcome: Change From Baseline to Week 26 in 6-minute Walk Distance (6MWD)
Description: The change from baseline to Week 26 in 6MWD was calculated as Week 26 minus baseline. The test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes. Missing values were imputed using a LOCF approach.
Time Frame: Baseline, Week 26
Population: Full analysis set included all randomized participants. Here, N (number of participants analyzed) signifies the number of participants analyzed for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: meter
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo)
Number analyzed (Participants) | 123 | 121
meter | 54.96 [40.419 to 69.501] | 56.39 [41.447 to 71.327]
Statistical Analysis 1: Comparison: Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) vs Double Oral Therapy (Macitentan, Tadalafil, and Placebo); Test type: Superiority; p = 0.8758, ANCOVA; Least Square (LS) Mean difference = -1.43, 95% CI 2-sided [-19.393 to 16.538]

3. Secondary Outcome: Change From Baseline to Week 26 in N-terminal Pro B-type Natriuretic Peptide (NT-proBNP) Levels
Description: The change from baseline to Week 26 in NT-proBNP was expressed as the ratio of Week 26 to baseline NT-proBNP (Week 26 divided by baseline). A geometric least square mean ratio of Week 26 to baseline NT-proBNP <1 corresponds to a reduction in NT-proBNP from baseline. Missing values were imputed using a LOCF approach.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ratio
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo)
Number analyzed (Participants) | 121 | 122
ratio | 0.26 [0.206 to 0.328] | 0.25 [0.200 to 0.320]
Statistical Analysis 1: Comparison: Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) vs Double Oral Therapy (Macitentan, Tadalafil, and Placebo); Test type: Superiority; p = 0.8529, ANCOVA; Ratio of geometric LS mean = 1.03, 95% CI 2-sided [0.770 to 1.371]

4. Secondary Outcome: Percentage of Participants With Absence of Worsening From Baseline to Week 26 in World Health Organization (WHO) Functional Class (FC)
Description: WHO FC is a classification graded from Class I to IV which reflects disease severity based on symptoms. Worsening was defined as death or hospitalization due to PAH. Class I: No limitation of activity; Class II: slight limitation with ordinary activities; Class III: may not have symptoms at rest but greatly limited activities; Class IV: symptoms at rest and inability to carry out any physical activity without symptoms. Missing values were imputed using a LOCF approach.
Time Frame: Week 26
Population: FAS included all randomized participants. Here, N (number of participants analyzed) signifies number of participants analyzed for this outcome measure. Participants with WHO FC IV at baseline were excluded from this analysis as they could not shift to a worse category.
Measure: Number; unit: percentage of participants
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo)
Number analyzed (Participants) | 122 | 119
percentage of participants | 99.2 | 97.5

5. Secondary Outcome: Change From Baseline to Week 26 in Mean Pulmonary Arterial Pressure (mPAP)
Description: Change from baseline to Week 26 in mean Pulmonary Arterial Pressure (mPAP) was measured. The pulmonary artery pressure is a measure of the blood pressure found in the main pulmonary artery. Missing values were imputed using a LOCF approach.
Time Frame: Baseline, Week 26
Population: Full analysis set included all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters of mercury (mmHg)
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo)
Number analyzed (Participants) | 123 | 124
millimeters of mercury (mmHg) | -12.92 [-14.609 to -11.235] | -12.20 [-13.881 to -10.515]
Statistical Analysis 1: Comparison: Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) vs Double Oral Therapy (Macitentan, Tadalafil, and Placebo); Test type: Superiority; p = 0.4998, ANCOVA; LS Mean Difference = -0.72, 95% CI 2-sided [-2.834 to 1.386]

6. Secondary Outcome: Change From Baseline to Week 26 in Mean Right Atrial Pressure (mRAP)
Description: Change from baseline to Week 26 in mean Right Atrial Pressure (mRAP) was measured. Missing values were imputed using a LOCF approach.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo)
Number analyzed (Participants) | 123 | 123
mmHg | -1.78 [-2.512 to -1.045] | -1.69 [-2.429 to -0.955]
Statistical Analysis 1: Comparison: Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) vs Double Oral Therapy (Macitentan, Tadalafil, and Placebo); Test type: Superiority; p = 0.8528, ANCOVA; LS Mean Difference = -0.09, 95% CI 2-sided [-1.003 to 0.830]

7. Secondary Outcome: Change From Baseline to Week 26 in Total Pulmonary Resistance
Description: Change from baseline to Week 26 in total pulmonary resistance was measured. Total pulmonary resistance was calculated as mPAP/CO*80, where CO is cardiac output. Re-calculated values were used for analysis and missing values were imputed using a LOCF approach.
Time Frame: Baseline, Week 26
Population: Full analysis set included all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: dynes*second per centimeter^5
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo)
Number analyzed (Participants) | 123 | 124
dynes*second per centimeter^5 | -511.88 [-569.36 to -454.40] | -514.28 [-571.45 to -457.11]
Statistical Analysis 1: Comparison: Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) vs Double Oral Therapy (Macitentan, Tadalafil, and Placebo); Test type: Superiority; p = 0.9474, ANCOVA; LS Mean Difference = 2.40, 95% CI 2-sided [-69.368 to 74.178]

8. Secondary Outcome: Change From Baseline to Week 26 in Cardiac Index
Description: Change from baseline to Week 26 in cardiac index was measured. Cardiac index is the amount of blood pumped by the heart, per minute, per meter square of body surface area. Re-calculated values were used for analysis and missing values were imputed using a LOCF approach.
Time Frame: Baseline, Week 26
Population: Full analysis set included all randomized participants.
Measure: Least Squares Mean (95% Confidence Interval); unit: liters per minute per meter square
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo)
Number analyzed (Participants) | 123 | 124
liters per minute per meter square | 0.97 [0.814 to 1.130] | 0.84 [0.684 to 0.997]
Statistical Analysis 1: Comparison: Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) vs Double Oral Therapy (Macitentan, Tadalafil, and Placebo); Test type: Superiority; p = 0.1902, ANCOVA; LS Mean Difference = 0.13, 95% CI 2-sided [-0.066 to 0.328]

9. Secondary Outcome: Change From Baseline to Week 26 in Venous Oxygen Saturation (%)
Description: Change from baseline to Week 26 in venous oxygen saturation was measured. Missing values were imputed using a LOCF approach.
Time Frame: Baseline, Week 26
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of oxygen saturation
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo)
Number analyzed (Participants) | 120 | 118
percentage of oxygen saturation | 5.59 [4.370 to 6.801] | 6.79 [5.561 to 8.020]
Statistical Analysis 1: Comparison: Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) vs Double Oral Therapy (Macitentan, Tadalafil, and Placebo); Test type: Superiority; p = 0.1227, ANCOVA; LS Mean Difference = -1.20, 95% CI 2-sided [-2.737 to 0.327]

10. Secondary Outcome: Number of Participants With Disease Progression Event
Description: Number of participants with disease progression event were reported. Disease progression event as adjudicated by the CEC, defined as any of the following: a. Death (all causes; adjudicated for PAH relationship); b. Hospitalization for worsening PAH; c. Initiation of prostacyclin, a prostacyclin analog, or a prostacyclin receptor agonist for worsening PAH; d. Clinical worsening defined as a post-baseline decrease in 6MWD by more than (>) 15 percent (%) from the highest 6MWD obtained at or after baseline, accompanied by WHO FC III or IV (both conditions confirmed at two consecutive post-baseline visits separated by 1-21 days).
Time Frame: Week 26, Month 12, Month 18, Month 24, Month 30, and End of Analysis Period (up to 40 months)
Population: Full analysis set included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo)
Number analyzed (Participants) | 123 | 124
Participants
  Week 26 | 8 | 13
  Month 12 | 13 | 20
  Month 18 | 15 | 23
  Month 24 | 15 | 25
  Month 30 | 16 | 27
  End of Analysis Period (up to 40 months) | 16 | 27
Statistical Analysis 1: Comparison: Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) vs Double Oral Therapy (Macitentan, Tadalafil, and Placebo); Test type: Superiority; p = 0.0867, Log Rank; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.32 to 1.09]

ADVERSE EVENTS:
Time Frame: Up to 42 Months
Description: The Safety Set included all participants who received at least one dose of any of 3 study treatments (macitentan, tadalafil, and selexipag or placebo) (Triple oral therapy= 123 participants and Double oral therapy= 123 participants). Four participants in triple therapy group did not receive selexipag and were therefore allocated to the double therapy group for the safety analyses.
Arm/Group | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo)
All-Cause Mortality (participants affected / at risk) | 4/119 | 12/127
Serious Adverse Events (participants affected / at risk) | 58/119 | 48/127
Other Adverse Events (participants affected / at risk) | 118/119 | 119/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) (N=119) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo) (N=127)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 3 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Microcytic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 2
Atrial Flutter (Cardiac disorders) | 0 | 2
Cardiac Arrest (Cardiac disorders) | 0 | 2
Cardiac Failure Chronic (Cardiac disorders) | 1 | 0
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 | 1
Left Ventricular Failure (Cardiac disorders) | 2 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial Effusion (Cardiac disorders) | 2 | 3
Right Ventricular Failure (Cardiac disorders) | 6 | 8
Supraventricular Tachycardia (Cardiac disorders) | 1 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Gastrointestinal Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 | 0
Deafness Neurosensory (Ear and labyrinth disorders) | 0 | 1
Blindness (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Amyloidosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 | 2
Gastrointestinal Polyp Haemorrhage (Gastrointestinal disorders) | 1 | 0
Incarcerated Umbilical Hernia (Gastrointestinal disorders) | 1 | 0
Large Intestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Rectal Prolapse (Gastrointestinal disorders) | 0 | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Accidental Death (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 2 | 3
Oedema Peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 0 | 1
Sudden Cardiac Death (General disorders) | 0 | 1
Sudden Death (General disorders) | 0 | 1
Autoimmune Hepatitis (Hepatobiliary disorders) | 1 | 0
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 | 0
Hepatic Cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Liver Disorder (Hepatobiliary disorders) | 1 | 0
Allergy to Arthropod Sting (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 2
Device Related Infection (Infections and infestations) | 1 | 0
Escherichia Sepsis (Infections and infestations) | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 0
Osteomyelitis Chronic (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 8 | 4
Pneumonia Legionella (Infections and infestations) | 1 | 0
Pneumonia Pseudomonal (Infections and infestations) | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 3
Septic Shock (Infections and infestations) | 1 | 1
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 2
Urosepsis (Infections and infestations) | 1 | 0
Vascular Device Infection (Infections and infestations) | 1 | 0
Chest Injury (Injury, poisoning and procedural complications) | 0 | 1
Deep Vein Thrombosis Postoperative (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Procedural Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0
Blood Pressure Increased (Investigations) | 0 | 1
Catheterisation Cardiac (Investigations) | 1 | 0
Haemoglobin Decreased (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 1
Influenza A Virus Test Positive (Investigations) | 0 | 1
Liver Function Test Increased (Investigations) | 1 | 0
Rotavirus Test Positive (Investigations) | 1 | 0
Sleep Study (Investigations) | 1 | 0
Transaminases Increased (Investigations) | 1 | 0
Waist Circumference Increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest Wall Haematoma (Musculoskeletal and connective tissue disorders) | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Systemic Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous Cell Carcinoma of the Tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Embolic Stroke (Nervous system disorders) | 0 | 1
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 6
Device Dislocation (Product Issues) | 2 | 0
Confusional State (Psychiatric disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 1 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 3 | 1
Nephropathy Toxic (Renal and urinary disorders) | 0 | 1
Prerenal Failure (Renal and urinary disorders) | 0 | 1
Renal Amyloidosis (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 1 | 0
Renal Impairment (Renal and urinary disorders) | 1 | 0
Scleroderma Renal Crisis (Renal and urinary disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Priapism (Reproductive system and breast disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Veno-Occlusive Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Respiratory Arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Drug Delivery Device Implantation (Surgical and medical procedures) | 1 | 1
Hip Arthroplasty (Surgical and medical procedures) | 1 | 2
Knee Arthroplasty (Surgical and medical procedures) | 0 | 1
Lung Transplant (Surgical and medical procedures) | 0 | 1
Open Reduction of Fracture (Surgical and medical procedures) | 1 | 0
Penile Operation (Surgical and medical procedures) | 1 | 0
Pericardial Drainage (Surgical and medical procedures) | 0 | 1
Therapy Change (Surgical and medical procedures) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 2
Hypertensive Crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 2
Paradoxical Embolism (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Acute Left Ventricular Failure (Cardiac disorders) | 1 | 0
Acute Right Ventricular Failure (Cardiac disorders) | 1 | 0
Atrial Tachycardia (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 1
Cardiac Failure Acute (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 1
Cardiac Failure High Output (Cardiac disorders) | 1 | 0
Cardiogenic Shock (Cardiac disorders) | 1 | 0
Coronary Artery Disease (Cardiac disorders) | 0 | 2
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Intestinal Ischaemia (Gastrointestinal disorders) | 1 | 0
Oesophageal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 1
Cardiac Electrophysiologic Study (Investigations) | 1 | 0
Transplant Evaluation (Investigations) | 0 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Carcinoma Cell Type Unspecified Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Toe Amputation (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Shock Haemorrhagic (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Triple Oral Therapy (Macitentan, Tadalafil, and Selexipag) (N=119) | Double Oral Therapy (Macitentan, Tadalafil, and Placebo) (N=127)
Anaemia (Blood and lymphatic system disorders) | 14 | 11
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 6 | 5
Palpitations (Cardiac disorders) | 14 | 11
Abdominal Distension (Gastrointestinal disorders) | 6 | 4
Abdominal Pain (Gastrointestinal disorders) | 7 | 6
Abdominal Pain Upper (Gastrointestinal disorders) | 8 | 7
Constipation (Gastrointestinal disorders) | 7 | 9
Diarrhoea (Gastrointestinal disorders) | 66 | 41
Dyspepsia (Gastrointestinal disorders) | 27 | 17
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 11 | 18
Nausea (Gastrointestinal disorders) | 56 | 33
Vomiting (Gastrointestinal disorders) | 30 | 14
Chest Discomfort (General disorders) | 7 | 10
Chest Pain (General disorders) | 6 | 4
Chills (General disorders) | 7 | 2
Fatigue (General disorders) | 24 | 22
Non-Cardiac Chest Pain (General disorders) | 10 | 6
Oedema Peripheral (General disorders) | 45 | 46
Pain (General disorders) | 11 | 9
Peripheral Swelling (General disorders) | 11 | 4
Pyrexia (General disorders) | 11 | 11
Bronchitis (Infections and infestations) | 6 | 6
Influenza (Infections and infestations) | 6 | 7
Nasopharyngitis (Infections and infestations) | 20 | 23
Upper Respiratory Tract Infection (Infections and infestations) | 14 | 21
Urinary Tract Infection (Infections and infestations) | 9 | 11
Alanine Aminotransferase Increased (Investigations) | 8 | 4
Aspartate Aminotransferase Increased (Investigations) | 10 | 4
Haemoglobin Decreased (Investigations) | 10 | 6
Weight Increased (Investigations) | 5 | 8
Decreased Appetite (Metabolism and nutrition disorders) | 14 | 4
Fluid Retention (Metabolism and nutrition disorders) | 6 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 17 | 15
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 19
Back Pain (Musculoskeletal and connective tissue disorders) | 13 | 19
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 9 | 7
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 8 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 21 | 19
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 37 | 24
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 35 | 15
Dizziness (Nervous system disorders) | 17 | 27
Headache (Nervous system disorders) | 83 | 78
Hypoaesthesia (Nervous system disorders) | 6 | 1
Paraesthesia (Nervous system disorders) | 8 | 2
Anxiety (Psychiatric disorders) | 9 | 5
Insomnia (Psychiatric disorders) | 8 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 25
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 13 | 13
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 22 | 23
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Pulmonary Arterial Hypertension (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Rash (Skin and subcutaneous tissue disorders) | 6 | 9
Swelling Face (Skin and subcutaneous tissue disorders) | 8 | 2
Flushing (Vascular disorders) | 21 | 22
Hypotension (Vascular disorders) | 10 | 8
Influenza Like Illness (General disorders) | 6 | 7
Sinusitis (Infections and infestations) | 5 | 8
Iron Deficiency (Metabolism and nutrition disorders) | 3 | 7

LIMITATIONS AND CAVEATS:
The main limitation of the sponsor's findings was that analyses of disease progression and mortality were exploratory due to the testing hierarchy and the post hoc nature of the analyses. The study was not powered to show significant differences for the disease progression related endpoint. Another limitation was the availability of hemodynamic assessments only for Week 26 timepoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation. Upon review, Actelion may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights.

DOCUMENTS (2):
  • Study Protocol (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/31/NCT02558231/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT02558231/SAP_002.pdf